CLINICAL TRIAL: NCT01602809
Title: Microvascular and Cardiac Dysfunction in Sickle Cell Disease
Brief Title: Microvessels and Heart Problems in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120124; 12-H-0124
Record Dates: First submitted 2012-05-18; First posted 2012-05-21 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10-25

CONDITIONS: Sickle Cell Disease
Keywords: Perfusion; Microvessels; Ultrasound; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Small blood vessels (microvessels) in many different organs are affected by diseases such as diabetes and atherosclerosis. These microvessels may also be abnormal in people who have sickle cell disease. Stiffness of the red blood cells leads to problems in the microvessels of the heart and kidneys. However, these problems may not be detected until these organs are severely affected. Researchers want to study problems with microvessels in people with and without sickle cell disease.

Objectives:

- To study how microvessels in the heart and other organs are affected by sickle cell disease.

Eligibility:

* Individuals at least 18 years of age who have sickle cell disease.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* All participants will have about 3 to 4 hours of testing for the study. Participants with sickle cell disease who are having a pain crisis at the time they enter the study may be asked to have the testing again when the crisis is over. The repeat testing will occur at least 4 weeks after the pain crisis ends.
* All participants will have the following tests:
* Blood draws to check kidney and liver function, and other blood tests
* Measure of blood flow in the brachial (upper arm) artery
* Heart ultrasound
* Ultrasound scans of arm muscles to study blood flow
* Ultrasound scans after taking vasodilators to increase blood flow
* Healthy volunteers will also have a magnetic resonance imaging scan. It will show blood flow in the heart. This scan will involve another dose of a vasodilator.

DETAILED DESCRIPTION:
Sickle cell disease is the most common genetic disease affecting African-Americans. It is characterized by an abnormal hemoglobin S, which polymerizes when deoxygenated leading to red cell rigidity and microvascular flow obstruction. Recurrent episodes of ischemia and a chronic inflammatory state lead to ischemia-reperfusion injury in multiple vital organ systems. Endothelial dysfunction has been demonstrated in patients with sickle cell disease and new therapies are targeted specifically towards the endothelium. Contrast ultrasound is a non-invasive technique that has been used to assess microvascular flow in coronary artery disease, diabetes, and other disease states. We propose to use this technique in sickle cell patients to compare their myocardial and skeletal muscle flow with that of normal controls, to detect changes during pain crisis, and to compare flow abnormalities with cardiac functional abnormalities.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult subject age greater than or equal to 18 years
* Able to give written informed consent
* For SCD groups, must have confirmed diagnosis of sickle cell disease

EXCLUSION CRITERIA:

* Atrial fibrillation or other irregular rhythm that would preclude adequate image acquisition
* Subjects with a contraindication for the ultrasound contrast agent.
* Pregnant or lactating women
* Known obstructive coronary or peripheral vascular disease
* SCD subjects at steady-state must not have acute pain crisis requiring intravenous analgesics within the prior 4 weeks
* SCD subjects in crisis must be within 72 hours of hospital admission
* Subjects with contraindications to MRI scanning will complete all other procedures but will not undergo the MRI scan. Subjects with an estimated glomerular filtration rate of <30 ml/min/1.73 m(2) will not receive gadolinium as per 2011 NHLBI gadolinium administration policy.
* Subjects with a contraindication to regadenson
* Any condition that in the clinical opinion of the investigators renders study procedures inadvisable.

Diagnosis of acute chest syndrome is not an exclusion criteria for this protocol. Subjects may be concurrently enrolled in any other protocols with the exception of investigational new drug studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-04-30; Study Completion 2017-10-25

PRIMARY OUTCOMES:
To use contrast-enhanced ultrasound to evaluate microvascular blood flow (MBF) and capillary RBC velocity (CBV) in skeletal muscle and the heart (at rest and during vasodilator stress) in patients with SCD in comparison to normal control patient...

SECONDARY OUTCOMES:
To determine whether MBF and CBV worsen during pain crisis in patients with SCD
To determine the relation between MBF and CBV and brachial artery flow or LV dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Sachdev, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kato GJ, Hebbel RP, Steinberg MH, Gladwin MT. Vasculopathy in sickle cell disease: Biology, pathophysiology, genetics, translational medicine, and new research directions. Am J Hematol. 2009 Sep;84(9):618-25. doi: 10.1002/ajh.21475. PMID 19610078
- [Background] Hebbel RP, Osarogiagbon R, Kaul D. The endothelial biology of sickle cell disease: inflammation and a chronic vasculopathy. Microcirculation. 2004 Mar;11(2):129-51. PMID 15280088
- [Background] Morris CR, Kuypers FA, Larkin S, Vichinsky EP, Styles LA. Patterns of arginine and nitric oxide in patients with sickle cell disease with vaso-occlusive crisis and acute chest syndrome. J Pediatr Hematol Oncol. 2000 Nov-Dec;22(6):515-20. doi: 10.1097/00043426-200011000-00009. PMID 11132219
- [Derived] Sachdev V, Sidenko S, Wu MD, Minniti CP, Hannoush H, Brenneman CL, Waclawiw MA, Arai AE, Schechter AN, Kato GJ, Lindner JR. Skeletal and myocardial microvascular blood flow in hydroxycarbamide-treated patients with sickle cell disease. Br J Haematol. 2017 Nov;179(4):648-656. doi: 10.1111/bjh.14918. Epub 2017 Sep 7. PMID 28880374